CLINICAL TRIAL: NCT04458168
Title: Feasibility and Evaluation of a Self-care App to Enhance Purposeful Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Rogel Cancer Center Cancer Control and Population Sciences O-SURE initiative (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2018.153; HUM00140226 (Other: University of Michigan)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recently completed treatment (Experimental): 25 women who have just completed treatment
  Interventions: Behavioral: Use of Purposeful app
- No recurrence of ovarian cancer for at least one year (Experimental): 25 women who have not experienced a recurrence of their ovarian cancer at least one year after their initial diagnosis
  Interventions: Behavioral: Use of Purposeful app
- Recurrence of ovarian cancer (Experimental): 25 women who have experienced a recurrence of their ovarian cancer after primary treatment
  Interventions: Behavioral: Use of Purposeful app

INTERVENTIONS:
Behavioral: Use of Purposeful app — Patients will be asked to use the Purposeful app every day, which should take no longer than 5 minutes. The app includes three key components: Explore, Act and Reflect. The Explore section provides thematically organized resources that suggest discrete actions users can try out and potentially incorporate into their lives. The app uses machine learning to customize resources presented to the user. The Act section is where users place actions they'd like to keep track of or build into a habit. Finally, the Reflect section includes daily "reflections" where the patient answers open ended questions regarding their alignment with their best self qualities, their sense of purpose, and more. Depending on whether users choose to allow push notifications, they will be notified daily to complete morning, afternoon, and/or evening reflections.
  Participants will complete questionnaires at enrollment and at 1, 3, and 6 months after enrollment.

SUMMARY:
In this pilot study, ovarian cancer survivors will be enrolled and followed for six months to evaluate usage of an eHealth app called "Purposeful".

DETAILED DESCRIPTION:
This study will determine the feasibility and acceptability of Purposeful, the eHealth app. First, feasibility of enrolling ovarian cancer survivors to use Purposeful will be assessed. Secondly, the acceptability of the app among ovarian cancer survivors will be assessed, based on frequency of use and validated acceptability measures. Participants will be asked to complete other validated questionnaires so investigators may explore whether further research on the Purposeful app among ovarian cancer survivors is warranted. This will include correlations between use of the Purposeful app and the life purpose questionnaire score. Lastly, correlation between life purpose and quality of life in ovarian cancer survivors will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian cancer or treatment for ovarian cancer through the University of Michigan Gynecologic Oncology service
* Completed primary treatment (either surgery alone or surgery + chemotherapy)
* Ability to understand and the willingness to sign a written informed consent
* Ability to speak and read English

Exclusion Criteria:

* There are no additional exclusion criteria for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by enrollment rate | At time of enrollment
  The number of patients who enroll in the study, of the total number of patients approached for enrollment.
Feasibility assessed by percentage of days of app use | 6 months
  Percentage of days during a 6-month period on which each participant used the Purposeful app. Using the app during the day is defined as doing at least one of the following: setting an intention; completing a reflection; completing an action. Usage data will be provided by the Purposeful app.
Feasibility assessed by trajectory of usage on a percent of days used on both a weekly and monthly time scale. | 6 months
  The average percentage of days of app use per week and per month during a 6-month period. Using the app during the day is defined as doing at least one of the following: setting an intention; completing a reflection; completing an action. Usage data will be provided by the Purposeful app.
Acceptability assessed by percentage of patients who find the Purposeful app to be acceptable | 6 months
  A score of 3 or more on the acceptability summary score (assessed using a protocol-specific questionnaire) will indicate that the patient finds the Purposeful app to be acceptable.

SECONDARY OUTCOMES:
Change in life purpose from baseline | 6 months
  Assessed at baseline, 1, 3 and 6 months using the Modified Ryff and Keyes Scales of Psychological Well-being evaluation, a 7-item questionnaire that uses a Likert scale ranging from 1 to 6, with higher scores indicating greater purpose in life.
Change in quality of life assessed using Functional Assessment of Cancer Therapy-Ovarian (FACT-O) Trial Outcome Index (TOI) (FACT-O TOI) | 6 months
  Assessed at baseline, 1, 3 and 6 months. FACT-O TOI is a 26-item questionnaire that sums the physical well-being, functional well-being, and additional health concerns with a 7-day recall period. All items will be rated on a 5 items (point) Likert Scale, from 0 (not at all) to 4 (very much so). To score the FACT-O TOI, all 26 items will be summed to create a single score with a range from 0 to 104. Items will be reverse scored when appropriate to provide a scale in which a higher score represent a higher quality of life.
Change in quality of life assessed using Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | 6 months
  Assessed at baseline, 1, 3 and 6 months. The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue with a 7-day recall period. All items will be rated on a 5 items (point) Likert Scale, from 0 (not at all) to 4 (very much so). To score the FACIT-fatigue, all 13 items will be summed to create a single fatigue score with a range from 0 to 52. Items will be reverse scored when appropriate to provide a scale in which a higher score represent less fatigue.
Change in quality of life using Comprehensive Measure of Meaning (Well-being questionnaire Part 10) | 6 months
  Assessed at baseline, 1, 3 and 6 months. The Comprehensive Measure of Meaning (Well-being questionnaire Part 10) is a 21-item questionnaire that uses a Likert scale ranging from 1 to 7, with higher scores indicating greater well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Leigh Pearce, PhD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States